CLINICAL TRIAL: NCT02667951
Title: Establishment and Effectiveness of a Community-based Long-term Care Model for Elderly Persons With Dementia
Brief Title: A Home-based Training Program for Elderly Patients With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yea-Ing Lotus Shyu, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSC 97-2420-H-182-002-MY3
Record Dates: First submitted 2016-01-23; First posted 2016-01-29 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Dementia
Keywords: Elderly; Dementia; Intervention program
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Caregivers received general information on dementia care and follow-up phone calls simply to maintain contact, but without any training for developing a behavioral problem-management plan and strategies.
- Intervention group (Experimental): Caregivers received solutions for managing behavioral problems, with referrals to community services and telephone consultation, further assurance and consultation were provided in monthly telephone follow-ups, and progress in behavior management was evaluated.
  Interventions: Other: A home-based caregiver-training program

INTERVENTIONS:
Other: A home-based caregiver-training program — A home-based caregiver-training program consisted of two weekly sessions, each lasting 2 to 3 hours. Following the training sessions, further assurance and consultation were provided in monthly telephone follow-ups, and progress in behavior management was evaluated.
  Arms: Intervention group

SUMMARY:
The illness course and symptoms of dementia is usually very long and characterized with behavioral, psychological and physical changes. Family caregivers' stresses change during the illness trajectory as well. The purpose of this study is to compare the costs and effectiveness of two care models- home-based caregiver-training program model and routine care model for dementia elders in Taiwan.

DETAILED DESCRIPTION:
The illness course and symptoms of dementia is usually very long and characterized with behavioral, psychological and physical changes. Family caregivers' stresses change during the illness trajectory as well. Thus, the needs of the elderly persons with dementia and their family caregivers differ in different stage of dementia, and the services they require are multidimensional. According to the researchers' previous 2-year study, behavioral problem management and service utilization were found to be the most difficult and least prepared caregiving activities and the family caregiver's needs for assistance of these two caregiving activities differed in different stage of dementia.The purpose of this study is to compare the costs and effectiveness of two care models- home-based caregiver-training program model and routine care model for dementia elders in Taiwan.

ELIGIBILITY:
Inclusion Criteria:(patients)

* diagnosed with dementia by a psychiatrist or neurologist
* Age 65 years or older
* living in a community of northern Taiwan
* living in a home setting
* scored >50 on the Chinese version Cohen-Mansfield Agitation Inventory (CMAI).

Exclusion Criteria:(patients)

* diagnosed with critical illness.

Inclusion Criteria:(caregivers)

* Primary caregiving responsibility and be at least 20 years old.

Exclusion Criteria:(caregivers)

* diagnosed with critical illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo LM, Huang HL, Liang J, Kwok YT, Hsu WC, Liu CY, Shyu YL. Trajectories of health-related quality of life among family caregivers of individuals with dementia: A home-based caregiver-training program matters. Geriatr Nurs. 2017 Mar-Apr;38(2):124-132. doi: 10.1016/j.gerinurse.2016.08.017. Epub 2016 Oct 6. PMID 27720499
- [Derived] Kuo LM, Huang HL, Liang J, Kwok YT, Hsu WC, Su PL, Shyu YL. A randomized controlled trial of a home-based training programme to decrease depression in family caregivers of persons with dementia. J Adv Nurs. 2017 Mar;73(3):585-598. doi: 10.1111/jan.13157. Epub 2016 Oct 17. PMID 27653753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 66 | 63
Completed | 45 | 40
Not Completed | 21 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 47 | 95
  >=65 years | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: year] | 56 (12) | 55 (15) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 14 | 62
  Male | 18 | 49 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Caregivers' Self-efficacy
Description: The Agitation Management Self-efficacy Scale was used to measure caregivers' self-efficacy for managing dementia patients' agitation. Caregivers were asked how confident they were about handling the problem for each identified behavioral problem and if they believed that they could manage the problem for behaviors that did not occur. Scores range from 42 to 210, with higher scores representing greater caregiver self-efficacy. In this study, Cronbach's alphas ranged from 0.98 to 0.99 at different time points.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale | 155 (34) | 178 (26)

2. Primary Outcome: Caregivers' Preparedness
Description: Preparedness was measured by the 10-item Caregiver Preparedness Scale,asks caregivers to rate how well prepared they think they are for seven domains of caregiving. A final question asks for an overall rating of how well prepared caregivers think they are to care for the care receiver. Items are scored on a 5-point Likert scale from 1 (not prepared) to 5 (well prepared). Scores range from 10 to 50, with higher scores representing greater preparedness for caregiving tasks. Validity and reliability of the original Preparedness scale was supported.24 The content validity index for the Preparedness Scale Taiwanese version was 1.0 and Cronbach's alpha for this scale among Taiwanese caregivers was 0.87. Cronbach's alpha in this study was 0.92.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale | 33 (8) | 38 (6)

3. Primary Outcome: Caregivers' Competence
Description: A 17-item Competence Scale was used to assess caregivers' knowledge and skills for managing behavioral problems of patients with dementia. Scores range from 17 to 85, with higher scores representing better competence. In this study, Cronbach's alpha ranged from 0.90 to 0.93 at different time points.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale | 51 (13) | 66 (8)

4. Primary Outcome: Dementia Patients' Behavioral Problems
Description: Physically aggressive behaviors of dementia patients were measured by the PAB subscale of the Chinese version CMAI, community form, which was shown to be valid and reliable for a Taiwanese sample. Each item (behavioral problem) is scored according to its frequency from 1 (never happens) to 7 (several times per hour). PAB subscale scores range from 7 to 49, with higher scores indicating more physically aggressive behaviors. In this study, the PAB subscale had Cronbach's alpha of 0.55.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale | 7.89 (1.66) | 7.88 (1.91)

5. Secondary Outcome: Caregivers' Quality of Life
Description: The Taiwan version of the Medical Outcomes SF-36 was used to measure family caregivers' HRQoL. The SF-36 contains eight generic health concepts: physical functioning (PF), role disability due to physical health problems (RP); bodily pain (BP); vitality (energy/fatigue) (VT); general health perceptions (GH); role disability due to emotional problems (RE); social functioning (SF); and general mental health (MH). Taiwan-specific SF-36 algorithms were used to compute the Mental Component Summary (MCS) and Physical Component Summary (PCS) scores using norm-based (mean = 50, SD = 10) scoring methods. Scores for each scale range from 0 to 100, with higher scores representing better health outcomes. In this study, Cronbach's alphas for the eight scales ranged from 0.81 to 0.99.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale
  PF | 80.22 (23.48) | 83.38 (26.00)
  RP | 67.22 (47.02) | 73.13 (43.63)
  RE | 70.37 (45.07) | 88.33 (29.77)
  SF | 68.06 (28.27) | 87.50 (17.68)
  BP | 72.84 (25.09) | 82.25 (18.75)
  VT | 52.00 (21.52) | 69.75 (13.77)
  MH | 64.09 (21.65) | 72.50 (13.07)
  GH | 50.64 (27.43) | 63.75 (22.22)
  PCS | 51.39 (9.72) | 52.96 (10.64)
  MCS | 50.10 (10.92) | 57.85 (7.11)

6. Secondary Outcome: Caregivers' Depressive Symptoms
Description: as for outcome 3
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 40
units on a scale | 13 (12) | 8 (7)

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/66 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No